CLINICAL TRIAL: NCT05995444
Title: A Phase 1, Single-Dose, Randomized, Placebo- and Positive-Control, Four-Way, Crossover Study for the Evaluation of the Effect of Epetraborole on QT Intervals in Healthy Adult Subjects
Brief Title: A Study to Assess the Effects of Epetraborole on the QT Interval in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AN2 Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EBO-104
Record Dates: First submitted 2023-06-27; First posted 2023-08-16 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers
Keywords: QTc; Epetraborole
MeSH Terms: interventions — Therapeutics; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Screening of subjects will occur within 28 days prior to the first dosing. Subjects will be housed on Day -1, at the time indicated by the CRU, until completion of study procedures on Day 2 of each period. On Day 1 of each period, subjects will receive 1 of 4 treatments: a single therapeutic dose of epetraborole (Treatment A), a single supratherapeutic dose of epetraborole (Treatment B), a single dose of epetraborole matching-placebo (Treatment C), or a single dose of moxifloxacin (Treatment D). Cardiodynamic ECGs and PK blood samples for epetraborole, metabolite M3, and moxifloxacin (as applicable) will be collected predose and for 24 hours postdose in each period. There will be a washout of at least 10 days between doses. Safety will be monitored throughout the study by repeated clinical and laboratory evaluations, including a follow-up visit approximately 14 days after the last dose.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 500 mg epetraborole (Experimental): 500 mg epetraborole
  Interventions: Drug: Epetraborole
- 2000 mg epetraborole (Experimental): 2000 mg epetraborole
  Interventions: Drug: Epetraborole
- Epetraborole-matching placebo (Placebo Comparator): Epetraborole-matching placebo
  Interventions: Drug: Epetraborole and matching placebo; Drug: Placebo
- 400 mg moxifloxacin (Active Comparator): 400 mg moxifloxacin
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Epetraborole and matching placebo — Treatment A (Therapeutic): 500 mg epetraborole (2 x 250 mg tablets) and epetraborole matching-placebo (6 tablets)
  Other Names: Therapeutic
  Arms: Epetraborole-matching placebo
Drug: Epetraborole — Treatment B (Supratherapeutic): 2000 mg epetraborole (8 x 250 mg tablets)
  Other Names: Supratherapeutic
  Arms: 2000 mg epetraborole; 500 mg epetraborole
Drug: Placebo — Treatment C (Placebo control): Epetraborole matching-placebo (8 tablets)
  Other Names: Placebo Control
  Arms: Epetraborole-matching placebo
Drug: Moxifloxacin — Treatment D (Positive control): 400 mg moxifloxacin (1 x 400 mg tablet)
  Other Names: Positive Control
  Arms: 400 mg moxifloxacin

SUMMARY:
A single-center, 4-way crossover study to evaluate the effect of single therapeutic and supratherapeutic oral doses of epetraborole on the heart rate (HR) corrected QT interval (QTc) by assessing concentration-QT (C-QT) relationship using exposure-response modeling.

DETAILED DESCRIPTION:
On Day 1 of each period, subjects will receive 1 of 4 treatments: a single therapeutic dose of epetraborole (Treatment A), a single supratherapeutic dose of epetraborole (Treatment B), a single dose of epetraborole-matching placebo (Treatment C), or a single dose of moxifloxacin (Treatment D). Cardiodynamic ECGs and PK blood samples for epetraborole, metabolite M3, and moxifloxacin (as applicable) will be collected predose and for 24 hours postdose in each period.

There will be a washout of at least 10 days between doses.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Adult, male or female, 18-65 years of age, inclusive, at the screening visit.
2. Subjects must agree to follow protocol-specified contraception guidance
3. Continuous non smoker for at least 3 months prior to the first dosing based on subject self-reporting
4. Body mass index (BMI) 18.0 and 32.0 kg/m2 at the screening visit.
5. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, and vital signs, as deemed by the Investigator or designee.
6. No clinically significant history or presence of ECG findings as judged by the Investigator or designee at the screening visit and first check-in

Exclusion Criteria:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
3. Presence of bacterial infections requiring the use of antibiotic therapy within 3 months prior to the first dosing.
4. History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing.
5. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months prior to the first dosing.
6. History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds (e.g., fluoroquinolones, epetraborole excipients), or allergy to ECG electrode adhesive patches or adhesive dressings/medical tape.
7. History or presence of any of the following, deemed clinically significant by the Investigator or qualified designee:

   1. Ventricular pre-excitation syndrome (Wolff Parkinson White syndrome)
   2. Arrhythmia or history of arrhythmia requiring medical intervention
   3. Risk factors for TdP (e.g., heart failure, cardiomyopathy, family history of Long QT Syndrome, or sudden unexpected cardiac death at a young age)
   4. Sick sinus syndrome, second- or third-degree atrioventricular block, myocardial infarction, pulmonary congestion, symptomatic or significant cardiac arrhythmia, prolonged QTcF interval, or conduction abnormalities
8. Is lactating or has a positive pregnancy test at the screening visit or first check-in (females only).
9. Positive urine drug or alcohol results at the screening visit or first check-in.
10. Positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) at the screening visit.
11. Positive results for coronavirus disease 2019 (COVID-19) at first check-in.
12. Unable to refrain from or anticipates the use of any drugs, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning

14 days prior to the first dosing.

13. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing.

14. Donation of blood or blood products or significant blood loss within 56 days prior to the first dosing or plans to donate blood products through the follow-up contact.

15. Participation in another clinical study and received an investigational agent within 30 days or within 5 half-lives (if known), prior to the first dosing, whichever is longer. The 30-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Changes to QTc interval | Study Day -1 to Study Day 2
  Effect of epetraborole plasma concentrations on the QTc interval using linear mixed effect exposure-response modeling, including the predicted ddQTc at Cmax values corresponding to exposure levels of interest.

SECONDARY OUTCOMES:
Effect of epetraborole plasma concentrations on other ECG parameters on QTc | Study Day -1 to Study Day 2
  Measure the Effect of epetraborole plasma concentrations on other ECG parameters on QTc
Assay sensitivity | Study Day -1 to Study Day 2
  Assay sensitivity assessment with ddQTc at the geometric mean Cmax value predicted from a linear mixed effect model evaluating the relationship between QTc and moxifloxacin plasma concentrations (exposure-response modeling).
Analysis of dQTc | Study Day -1 to Study Day 2
  QTc interval using a mixed effect analysis of covariance (ANCOVA) carried out as appropriate to analyze dQTc at each time point post baseline.
PK Concentration analysis for epetraborole and metabolite M3 of AUC0 t | Study Day -1 to Study Day 2
  Analysis of PK Concentration for epetraborole and metabolite M3 of AUC0 t
Evaluation of TEAEs | Study Day 1 through Study Day 14
  TEAEs
Safety Vital Signs changes of body temperature | Study Day 1 through Study Day 14
  Measure Safety Vital Signs changes of body temperature
Orthostatic Vital Signs changes of Heart Rate from supine to standing position. | Study Day 1 through Study Day 14
  Measure Orthostatic Vital Signs changes of Heart Rate from supine to standing position.
Effect of epetraborole plasma concentrations on other ECG parameters on, PR | Study Day -1 to Study Day 2
  Measure the Effect of epetraborole plasma concentrations on other ECG parameters on, PR
Effect of epetraborole plasma concentrations on other ECG parameters on QRS duration | Study Day -1 to Study Day 2
  Measure the Effect of epetraborole plasma concentrations on other ECG parameters on QRS duration.
Effect of epetraborole plasma concentrations on other ECG parameters on HR. | Study Day -1 to Study Day 2
  Measure the Effect of epetraborole plasma concentrations on other ECG parameters on HR.
PK Concentration analysis for epetraborole and metabolite M3 of AUC0 inf | Study Day -1 to Study Day 2
  Analysis of PK Concentration for epetraborole and metabolite M3 of AUC0 inf
PK Concentration analysis for epetraborole and metabolite M3 of AUC%extrap | Study Day -1 to Study Day 2
  Analysis of PK Concentration for epetraborole and metabolite M3 of AUC%extrap
PK Concentration analysis for epetraborole and metabolite M3 of Cmax | Study Day -1 to Study Day 2
  Analysis of PK Concentration for epetraborole and metabolite M3 of Cmax
PK Concentration analysis for epetraborole and metabolite M3 of Tmax | Study Day -1 to Study Day 2
  Analysis of PK Concentration for epetraborole and metabolite M3 of Tmax
PK Concentration analysis for epetraborole and metabolite M3 of Kel | Study Day -1 to Study Day 2
  Analysis of PK Concentration for epetraborole and metabolite M3 of Kel
PK Concentration analysis for epetraborole and metabolite M3 of t½ | Study Day -1 to Study Day 2
  Analysis of PK Concentration for epetraborole and metabolite M3 of t½
PK Concentration analysis for epetraborole and metabolite M3 of CL/F (parent only), | Study Day -1 to Study Day 2
  Analysis of PK Concentration for epetraborole and metabolite M3 of CL/F (parent only),
PK Concentration analysis for epetraborole and metabolite M3 of Vz/F (parent only) | Study Day -1 to Study Day 2
  Analysis of PK Concentration for epetraborole and metabolite M3 of Vz/F (parent only
PK Concentration analysis for epetraborole and metabolite M3 of MR AUC0 t | Study Day -1 to Study Day 2
  Analysis of PK Concentration for epetraborole and metabolite M3 of MR AUC0 t
PK Concentration analysis for epetraborole and metabolite M3 of MR AUC0 inf | Study Day -1 to Study Day 2
  Analysis of PK Concentration for epetraborole and metabolite M3 of MR AUC0 inf
PK Concentration analysis for epetraborole and metabolite M3 of MR Cmax | Study Day -1 to Study Day 2
  Analysis of PK Concentration for epetraborole and metabolite M3 of MR Cmax
Safety Vital Signs changes of respiratory rate | Study Day 1 through Study Day 14
  Measure Safety Vital Signs changes of respiratory rate
Safety Vital Signs changes of blood pressure | Study Day 1 through Study Day 14
  Measure Safety Vital Signs changes of blood pressure (systolic and diastolic)
Safety Vital Signs changes of heart rate | Study Day 1 through Study Day 14
  measure Safety Vital Signs changes of heart rate
Orthostatic Vital Signs changes of blood pressure from supine to standing position. | Study Day 1 through Study Day 14
  Measure Orthostatic Vital Signs changes of blood pressure from supine to standing position (systolic and diastolic).

CONTACTS AND LOCATIONS:
Locations (1):
- 423001, Tempe, Arizona, United States